CLINICAL TRIAL: NCT07356050
Title: Verifying Antibodies After Live Immunization Delivery (VALID): a Study of Measles Vaccine Immunogenicity in Children With Sickle Cell Disease
Acronym: VALID
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Thrasher Research Fund (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: VALID
Record Dates: First submitted 2026-01-07; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease; Measles Vaccination; Sickle Cell Anemia
Keywords: Measles Vaccine Immunogenicity
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At maximum, 3 mL of whole blood will be collected from participants. Plasma will be separated from the whole blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Second Measles Vaccine (MV2): Participants who receive second measles vaccine.
- First Measles Vaccine (MV1): Participants who obtain the first measles vaccine.

SUMMARY:
The goal of this study is to learn if infants with sickle cell disease (SCD) develop adequate protection after measles vaccines. (not looking at any prolonged duration)

DETAILED DESCRIPTION:
Families of infants with SCD who are eligible for a measles vaccine per standard care will be contacted to discuss enrollment in the study. One cohort will be evaluated for response to the first measles vaccine (MV1) and another cohort will be evaluated for response to the second measles vaccine (MV2). Blood samples will be collected from participants prior to measles vaccination and then again at 4 and 8 weeks after vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with confirmed Sickle Cell Disease.
2. Participants 6 months and 6 years of age and due for measles vaccination within 3 months per national guidelines.
3. Willing and able to provide informed consent
4. Ability to comply with study related evaluations and follow-up visits.

Exclusion Criteria:

1. Known primary immunodeficiency syndrome, cancer, or acquired immunodeficiency syndrome (AIDS) that would preclude vaccination with live virus vaccines.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from 6 months to 6 years old with Sickle Cell Disease who receive medical care in Cincinnati, Ohio; Accra, Ghana; and Mwanza, Tanzania will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Measles Seroconversion Rates 8 Weeks After MV1 and MV2 Vaccinations | From enrollment to the end of sample collection at 8 weeks
  Sample analysis of 126 participants 8-weeks post complete measles vaccination.

SECONDARY OUTCOMES:
Measles Seroconversion Rates 4 Weeks After MV1 Vaccination | From enrollment to the end of sample collection at 4-weeks post first vaccination.
  Sample analysis of participants' seroconversion rates 4-weeks post first vaccination.
Measles Seroconversion Rates 4 Weeks after MV2 Vaccination | From second vaccination to end of sample collection at 4-weeks post second vaccination.
  The sample analysis of participant's seroconversion rates 4-weeks post second vaccination.
Variables Associated with Measles Vaccine-induced Antibody Response | From enrollment to the end of sample collection at 8 weeks.
  Identify participant's demographic, clinical history, and sickle cell treatments as variables to measles antibody response.
Modalities for Sample Analysis | Through study completion, an average of 12 weeks.
  Compare sample analysis results between the gold standard (serum or plasma) and Mitra sample using dried blood spot or whole blood.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Power-Hays, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States
- Korle Bu Teaching Hospital, Accra, Ghana, Ghana
- Bugando Medical Centre, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: No